CLINICAL TRIAL: NCT00244088
Title: Study of the Etiology of Intra-Abdominal Infections
Brief Title: Study Evaluating the Etiology of Intra-Abdominal Infections
Status: Completed | Type: Observational
Sponsor: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Other Study IDs: 101316
Record Dates: First submitted 2005-10-21; First posted 2005-10-25 (Estimated); Last update posted 2009-09-01 (Estimated); Status verified 2009-08

CONDITIONS: Intra-abdominal Infection
Keywords: Abdominal infection
MeSH Terms: conditions — Intraabdominal Infections

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Intra-abdominal fluid

SUMMARY:
The aim of this study is to define the etiology of intra-abdominal infections, to study the role of Enterococcus spp and Pseudomonas aeruginosa in these infections and to clarify the need for specific enterococcal antimicrobial coverage.

ELIGIBILITY:
Inclusion Criteria:

* A case will be defined as an intra-abdominal abscess or peritoneal fluid culture that will be positive for enterococcus or an enterococcal bacteriemia in association with an intra-abdominal source of infection.
* A control will be defined as a culture-positive intra-abdominal infection or bacteriemia due to an intraabdominal focus where enterococci have not been isolated.

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Surgery units
Sampling Method: Non-Probability Sample
Enrollment: 340
Dates: Start 2004-04; Primary Completion 2004-12 (Actual); Study Completion 2004-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Principal Investigator — Wyeth is now a wholly owned subsidiary of Pfizer